CLINICAL TRIAL: NCT03312036
Title: HEpatic Regeneration With COupled Plasma Filtration and Adsorption for Liver Extracorporeal Detoxification
Acronym: HERCOLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Gabriele Donati, M.D. PhD, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 87/2012/O/Disp
Record Dates: First submitted 2017-09-28; First posted 2017-10-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Liver Failure, Acute; Liver Failure, Acute on Chronic
Keywords: CPFA; Liver failure; Resin; detoxification
MeSH Terms: conditions — Liver Failure, Acute; Acute-On-Chronic Liver Failure; Liver Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CPFA Patients (Experimental): Patients affected by acute or acute on chronic liver failure who undergo Coupled plasma filtration and adsorption (CPFA) to recover their basal liver function or as a bridge to liver transplantation. The intervention is CPFA treatment which lasts 6 hour length. The intervention can be repeated for a maximum of 5 times.
  Interventions: Device: Coupled plasma filtration and adsorption (CPFA)

INTERVENTIONS:
Device: Coupled plasma filtration and adsorption (CPFA) — Patients affected by acute or acute on chronic liver failure are enrolled to undergo CPFA extracorporeal treatments and the standard medical therapy to recover their basal liver function or as a "bridge" to liver transplantation

SUMMARY:
CPFA is currently used in the treatment of severe sepsis with the intention of removing the proinflammatory mediators from the systemic circulation. Some evidence exists about the bilirubin adsorbing ability of the neutral styrenic resin which is part of the extracorporeal circuit of CPFA. The aim of this study is to assess efficacy and safety of CPFA in extracorporeal detoxification of liver toxins in patients affected by acute or acute-on-chronic liver failure.

DETAILED DESCRIPTION:
CPFA allows an improvement of blood pressure and inflammatory response during sepsis and multiorgan failure. This extracorporeal detoxification system was developed to non-specifically remove larger mediators during systemic inflammation with an extracorporeal circuit consisting of a plasma filter, a resin cartridge and a high-flux dialyzer. At present it is performed with the use of a five-pump modular treatment consisting of a plasma filter and a following absorption on an unselective hydrophobic resin cartridge and a final passage of the reconstituted blood through a high permeability polyethersulfone haemofilter, in which convective exchanges may be applied in a postdilution mode. Ronco et al. in 2002 compared CPFA treatment to continuous veno-venous haemodiafiltration (CVVHDF) in 10 patients affected by septic shock. The patients underwent 10-hour length CPFA and an increase of arterial blood pressure and a significant reduction of norepinephrine dosage were observed in comparison to the arterial blood pressure and the norepinephrine dosage achieved with the CVVHDF treatment. Formica et al. in 2004 confirmed these results using 100 CPFA treatments in 12 patients affected by septic shock with or without acute kidney injury. Patient survival at 28 days was 90%, while survival of after 90 days was 70%. Mao et al. also compared CPFA with High Volume Hemofiltration and they showed that CPFA increased the ratio between anti-inflammatory and pro-inflammatory cytokines; CPFA enhanced Human Leucocyte Antigen (HLA) class II expression on monocytes and improved the leukocyte response to inflammation measuring leukocyte production of Tumor Necrosis Factor-alfa. Recently Livigni et al. on behalf of the Italian group for the evaluation of interventions in intensive care medicine carried out a randomised controlled trial enrolled 330 adult patients with septic shock, 192 were randomised to either have CPFA added to the standard care, or not. CPFA was to be performed daily for 5 days, lasting at least 10 h/day. The trial was stopped because nearly 50% of the patients could not achieve treatment completion due to technical reasons (primarily coagulation). The trial did observe that patients with the highest amounts of treated plasma appeared to have a survival benefit. The technique underwent further modifications to improve the technical aspects and anticoagulation and a new trial is now underway with a high dose of plasma > 0.18 litres/ kg/ day.

As to the hepatic toxin removal it depends on the ability of the detoxification system to extract albumin bound toxins by means of adsorption. The adsorption consists in the consolidation on the surface of a solid material of molecules floating in a fluid after matching the fluid with the solid. The consolidation is due to weak bounds as in the case of Van der Waals and hydrophobic bounds. The selectivity of adsorption occurs when albumin molecules easily pass throughout the sorbent while the sorbent draw the albumin carried toxins into the pores of the sorbent. The hepatic toxins often are hydrophobic and with molecular weight < 1,000 daltons (bilirubin = 406 daltons, cholic acid = 283 daltons, chenodeoxycholic acid = 272 daltons). The albumin structure consists in 3 domains, which allows a multi-binding protein transport. As to bilirubin, its protein binding is a physiological protective mechanism to prevent the free bilirubin diffusion and toxicity in human tissues. The amount of bilirubin production is about 300 gr/day. The molecule most tightly bound to albumin is non-conjugated bilirubin: the amount of non-conjugated bilirubin not bound to albumin is < 0.1%. Non-conjugated bilirubin is currently considered as "indirect" bilirubin because it gives an indirect reaction with standard diazo reagents. Conjugated bilirubin is also bound to albumin but with a reduced affinity. The albumin-bilirubin bond occurs by means of covalent or non-covalent strengths. The 2 bilirubin binding sites on albumin show different constant of association (Ka). The primary site has a high affinity, its Ka is 55-68 micromol/L and it can bind only 1 mole of bilirubin. The secondary site has a low affinity, its Ka is 4.4-5.0 micromol/L and it can bind more than 1 mole of bilirubin. A gap between 20 and 50 ångström between albumin and the sorbent is needed to move bilirubin from albumin to the sorbent.

The CPFA efficacy on bilirubin adsorption is based on hydrophobic polystyrene-divinylbenzene copolymer matrices of the resin cartridge that have mean pore sizes of 30 nanometres. Harm et al. reported that the hydrophobic polystyrene-divinylbenzene copolymer of CPFA resin cartridge (type B copolymer: mean diameter 128 micron, pore size 30 nanometres and surface area of 700 m2/gr of resin) binds higher amount of bilirubin than the amount of bilirubin bound with the other kinds of polystyrene-divinylbenzene copolymer matrices tested (type A copolymer: mean diameter 120 micron, pore size 15 nanometres and surface area of 900 m2/gr of resin; type C copolymer: mean diameter 37 micron, pore size 100 nanometres and surface area of 200 m2/gr of resin).

Few authors in vivo assessed the bilirubin adsorbing ability of the neutral styrenic resin of CPFA. Caroleo et al. reported the first case of hepatic toxins removal by means of CPFA in a patient affected by acute liver failure due to cardiogenic shock. Maggi et al. reported 2 further cases where bilirubin removal was obtained in 2 patients with delayed graft function after liver transplantation. The patients achieved a 40% bilirubin reduction after 3 treatments with CPFA lasting 3-hours each.

ELIGIBILITY:
Inclusion Criteria:

* Acute liver failure
* Acute on chronic liver failure
* Bridge to liver transplantation

Exclusion Criteria:

* acute hemorrhage
* shock
* respiratory failure
* acute coronary syndrome
* psychiatric illnesses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-06-06 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
The mortality reduction of patients with acute or acute on chronic liver failure; | 1 year
  The measure is the overall survival of the patients after CPFA and standard medical therapy

SECONDARY OUTCOMES:
Efficacy of liver toxins detoxification | 1 year.
  The measures of efficacy consist in the evaluation bilirubin levels, biliary acids levels, ammonia levels and lactate levels
Improvement of hepatic encephalopathy | 1 year
  The measure of hepatic encephalopathy is assessed by means of the West Haven Criteria
Improvement of the arterial blood pressure of the patients | 1 year
  Measuring arterial blood pressure (mmHg) on starting CPFA, during the CPFA treatment and at CPFA end.
Biocompatibility of CPFA | 1 year
  Blood leukocytes, platelets, Hemoglobin are assessed before and after each CPFA treatment
Cytokines clearance during CPFA | 1 year
  Interleukin-6, Tumor Necrosis Factor alfa, Interleukin-10, Hepatocyte growth factor are assessed before and after each CPFA treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano La Manna, Prof., Principal Investigator — University of Bologna
Locations (1):
- Nephrology Dialysis and Renal Transplantation Unit, S.Orsola University Hospital, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ronco C, Brendolan A, d'Intini V, Ricci Z, Wratten ML, Bellomo R. Coupled plasma filtration adsorption: rationale, technical development and early clinical experience. Blood Purif. 2003;21(6):409-16. doi: 10.1159/000073444. PMID 14586184
- [Background] Tetta C, Cavaillon JM, Schulze M, Ronco C, Ghezzi PM, Camussi G, Serra AM, Curti F, Lonnemann G. Removal of cytokines and activated complement components in an experimental model of continuous plasma filtration coupled with sorbent adsorption. Nephrol Dial Transplant. 1998 Jun;13(6):1458-64. doi: 10.1093/ndt/13.6.1458. PMID 9641176
- [Background] Cole L, Bellomo R, Davenport P, Tipping P, Uchino S, Tetta C, Ronco C. The effect of coupled haemofiltration and adsorption on inflammatory cytokines in an ex vivo model. Nephrol Dial Transplant. 2002 Nov;17(11):1950-6. doi: 10.1093/ndt/17.11.1950. PMID 12401852
- [Background] Ronco C, Brendolan A, Lonnemann G, Bellomo R, Piccinni P, Digito A, Dan M, Irone M, La Greca G, Inguaggiato P, Maggiore U, De Nitti C, Wratten ML, Ricci Z, Tetta C. A pilot study of coupled plasma filtration with adsorption in septic shock. Crit Care Med. 2002 Jun;30(6):1250-5. doi: 10.1097/00003246-200206000-00015. PMID 12072677
- [Background] Formica M, Olivieri C, Livigni S, Cesano G, Vallero A, Maio M, Tetta C. Hemodynamic response to coupled plasmafiltration-adsorption in human septic shock. Intensive Care Med. 2003 May;29(5):703-8. doi: 10.1007/s00134-003-1724-0. Epub 2003 Mar 29. PMID 12665998
- [Background] Mariano F, Tetta C, Stella M, Biolino P, Miletto A, Triolo G. Regional citrate anticoagulation in critically ill patients treated with plasma filtration and adsorption. Blood Purif. 2004;22(3):313-9. doi: 10.1159/000078788. PMID 15256798
- [Background] Lentini P, Cruz D, Nalesso F, de Cal M, Bobek I, Garzotto F, Zanella M, Brendolan A, Piccinni P, Ronco C. [A pilot study comparing pulse high volume hemofiltration (pHVHF) and coupled plasma filtration adsorption (CPFA) in septic shock patients]. G Ital Nefrol. 2009 Nov-Dec;26(6):695-703. Italian. PMID 19918752
- [Background] Mao HJ, Yu S, Yu XB, Zhang B, Zhang L, Xu XR, Wang XY, Xing CY. Effects of coupled plasma filtration adsorption on immune function of patients with multiple organ dysfunction syndrome. Int J Artif Organs. 2009 Jan;32(1):31-8. doi: 10.1177/039139880903200104. PMID 19241361
- [Background] Livigni S, Bertolini G, Rossi C, Ferrari F, Giardino M, Pozzato M, Remuzzi G; GiViTI: Gruppo Italiano per la Valutazione degli Interventi in Terapia Intensiva (Italian Group for the Evaluation of Interventions in Intensive Care Medicine) is an independent collaboration network of Italian Intensive Care units. Efficacy of coupled plasma filtration adsorption (CPFA) in patients with septic shock: a multicenter randomised controlled clinical trial. BMJ Open. 2014 Jan 8;4(1):e003536. doi: 10.1136/bmjopen-2013-003536. PMID 24401721
- [Background] Hughes RD. Review of methods to remove protein-bound substances in liver failure. Int J Artif Organs. 2002 Oct;25(10):911-7. doi: 10.1177/039139880202501003. PMID 12456030
- [Background] Weiss JS, Gautam A, Lauff JJ, Sundberg MW, Jatlow P, Boyer JL, Seligson D. The clinical importance of a protein-bound fraction of serum bilirubin in patients with hyperbilirubinemia. N Engl J Med. 1983 Jul 21;309(3):147-50. doi: 10.1056/NEJM198307213090305. PMID 6866015
- [Background] Gong D, Cruz D, Ronco C. Depurative capacity of molecular adsorbent recycling system (MARS): A focus on bilirubin removal. Int J Artif Organs. 2008 Oct;31(10):875-81. doi: 10.1177/039139880803101003. PMID 19009505
- [Background] Harm S, Falkenhagen D, Hartmann J. Pore size--a key property for selective toxin removal in blood purification. Int J Artif Organs. 2014 Sep;37(9):668-78. doi: 10.5301/ijao.5000354. Epub 2014 Sep 23. PMID 25262632
- [Background] Caroleo S, Rubino AS, Tropea F, Bruno O, Vuoto D, Amantea B, Renzulli A. Coupled plasma filtration adsorption reduces serum bilirubine in a case of acute hypoxic hepatitis secondary to cardiogenic shock. Int J Artif Organs. 2010 Oct;33(10):749-52. PMID 21058270
- [Background] Maggi U, Nita G, Gatti S, Antonelli B, Paolo R, Como G, Messa P, Rossi G. Hyperbilirubinemia after liver transplantation: the role of coupled plasma filtration adsorption. Transplant Proc. 2013 Sep;45(7):2715-7. doi: 10.1016/j.transproceed.2013.07.019. PMID 24034030